CLINICAL TRIAL: NCT05771246
Title: Third Molar Agenesis Related To Craniofacial Pattern And Sella Turcica Bridging: A Retrospective Cephalometric Study
Brief Title: Craniofacial Morphology And Sella Turcica Bridging Associated With Third Molar Agenesis.
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2023-AGENESISTHIRDMOLAR
Record Dates: First submitted 2023-02-17; First posted 2023-03-16 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Tooth Agenesis
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with third molar agenesis.
  Interventions: Diagnostic Test: Radiographic evaluation
- Control group: Patients with the presence of all third molars.
  Interventions: Diagnostic Test: Radiographic evaluation

INTERVENTIONS:
Diagnostic Test: Radiographic evaluation — Panoramic and lateral cephalometric radiographs with cephalometric analysis will be performed.

SUMMARY:
The aim of this retrospective study is to analyze the third molar agenesis with respect to sella turcica bridging and other craniofacial patterns in patients asking for orthodontic consultation. The main question[s] it aims to answer are:

* is there a relationship between third molar agenesis and sella turchina bridging?
* is there a relationship between third molar agenesis and craniofacial patterns?

DETAILED DESCRIPTION:
Patients referring for orthodontic consultation at the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic and Pediatric Sciences, University of Pavia, 27100 Pavia, Italy, will be enrolled for the study according to the inclusion criteria. For each patient, lateral cephalometric radiograph and panoramic radiograph will be performed. For each lateral cephalometric radiograph, a cephalometric tracing will be performed with DeltaDent software (version 2.5.12, Outside Format, Pandino, Italy). Riedel's ANB angle [Riedel 1952] has been chosen to determine patients' skeletal class. Steiner's SN^GoGn angle [Steiner 1953] has been chosen to evaluate skeletal divergence. Facial axis (BaNa^CCGn), Lower Facial Height (LFH) and mandibular plan angle (FH^GoMe) from Rickett's analysis [Rickett's 1961] have been adopted to determine facial growth. According to Jaraback's cephalometric analysis [Jaraback 1985], saddle angle, articular angle, upper gonial angle, lower gonial angle will be measured to assess the growth pattern. Linear measurements of sella depth, sella diameter and interclinoid distance [Silverman 1957; Kisling 1966] will be calculated. Linear regressions between craniofacial patterns, sella turcica bridging and third molar agenesis will be calculated. A control group with no third molar agenesis will be provided.

ELIGIBILITY:
Inclusion Criteria:

* G stage of Demirjian's classification for third molar maturation or absence of third molar germs
* Patients with one lateral cephalometric digital radiograph executed in Natural Head Position (patients were asked to keep the teeth in contact and the lips relaxed).
* Patients with panoramic radiograph;

Exclusion Criteria:

* Ascertained previous surgical extraction/s of third molar/s
* Orthopedic/orthodontic therapy
* Orthognathic surgery.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referring to the Unit of Orthodontics and Pediatric Dentistry for orthodontic consultation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Linear regression between third molar agenesis and ANB | Baseline
  ANB is calculated according to Riedel's analysis: angle formed between Point A (maxillary sovraspinal point), point B (Bubmental mandibular point) and N (Nasion)
Linear regression between third molar agenesis and Interclinoid Distance | Baseline
  Distance between tuberculum sella (TS) and dorsum sella (DS).
Linear regression between third molar agenesis and Sella Depth. | Baseline
  Distance of a line dropped perpendicular from the interclinoid distance to the deepest point of the sella floor.
Linear regression between third molar agenesis and Sella Diameter | Baseline
  Distance between tuberculum sella and the farthest point on the inner wall of the sella.
Linear regression between third molar agenesis and Sn^GoGn. | Baseline
  Steiner's Sn^GoGn is the angle formed between 2 planes: cranial base line (SN) and mandibular plane (GoGn)
Linear regression between third molar agenesis and ArGo^GoGn | Baseline
  Jaraback's Ar^Go^Gn is the angle formed between the 2 planes: ArGo and GoGn

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, Ms, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator